CLINICAL TRIAL: NCT06398665
Title: Image-guided, Accelerated, Theta-burst Stimulation for the Treatment of Post-concussion Syndrome - Open-label Pilot Study
Brief Title: Accelerated, Theta-burst Stimulation for the Treatment of Post-concussion Syndrome - Open-label Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Sean Michael Nestor, clinician-investigator and interventional psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6160
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Post-Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: This open-label pilot study aims to investigate the potential of a non-invasive brain stimulation technique, accelerated intermittent theta-burst stimulation (iTBS) repetitive transcranial magnetic stimulation (rTMS), for treating post- concussive syndrome (PCS) in persons with mild traumatic brain injury (mTBI).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated Intermittent Theta-Burst Stimulation (Experimental): Non-invasive brain stimulation technique, accelerated intermittent theta-burst stimulation (iTBS) repetitive transcranial magnetic stimulation (rTMS), for treating post- concussive syndrome (PCS) in persons with mild traumatic brain injury
  Interventions: Device: Intermittent Theta-Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta-Burst Stimulation — Accelerated course of left dlPFC iTBS, consisting of 600 pulses/session, 50 minutes intersession interval, 8 session/day for 5 days) at 90% resting motor threshold (MT)

SUMMARY:
The current study aims to better understand the efficacy of intermittent theta-burst stimulation (iTBS) treatment in patients diagnosed with post-concussion syndrome (PCS) and to explore changes in brain networks after undergoing iTBS to assess its safety and feasibility in treating PCS.

DETAILED DESCRIPTION:
This open-label pilot study aims to investigate the potential of a non-invasive brain stimulation technique, accelerated intermittent theta-burst stimulation (iTBS) repetitive transcranial magnetic stimulation (rTMS), for treating post- concussive syndrome (PCS) in persons with mild traumatic brain injury (mTBI). PCS is characterized by symptoms like cognitive impairment, mood dysregulation, fatigue, and headaches, with limited treatment options. Previous research has indicated brain network dysfunction in mTBI patients and suggested the potential of conventional once daily high frequency rTMS for treating PCS symptoms. Our proposal builds on these findings by utilizing the expertise and resources of Sunnybrook's Harquail Centre for Neuromodulation, which has extensive experience in delivering rTMS and theta-burst stimulation for treatment-resistant depression. This pilot study will implement an accelerated iTBS rTMS protocol, offering shorter treatment duration, as well as MRI-guided stimulation for precise targeting. The investigators will also explore changes in brain function following rTMS using a technique called functional magnetic resonance imaging. The investigators ultimately aim to understand how iTBS may alter the post-concussive brain and the extent to which these changes may improve PCS.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of head trauma sufficiently severe to result in loss of consciousness, post-traumatic amnesia and/or acute altered mental status.
* At least three symptoms including headache, dizziness, fatigue, irritability, insomnia, memory difficulties, concentration difficulties, mood dysregulation.
* Onset of symptoms within 4 weeks following the head trauma.
* Age 18-60, inclusive.
* Persistence of PCS symptoms for at least 3 months but less than 24 months
* Able to provide informed consent and comply with the study protocol
* Patients will not be excluded solely on the basis of communication (i.e., non-English speaking) unless they have exclusion criteria that is the cause of the communication difficulties.

Exclusion Criteria:

* Evidence of major structural neuroimaging abnormalities (e.g., intracranial hemorrhage, skull fracture or a large intracranial lesion)
* History of prior rTMS therapy,
* Contraindications to MRI (e.g., pacemaker, metallic implants etc.).
* Ferromagnetic, non-removable metallic implants from above the clavicle with the exception of dental work.
* Active personal injury litigation
* History of seizure disorder, not including febrile seizures in childhood
* Substance dependence within the last 6 months
* Pregnant
* Currently taking more than lorazepam 2 mg daily (or benzodiazepine equivalent) or any dose of an anticonvulsant (due to the potential to reduce rTMS efficacy)
* Currently taking an antiepileptic medication
* Mild and major comorbid medical conditions (as determined by investigators - e.g., neurological diseases, uncontrolled hypertension or diabetes, malignancy)
* A major comorbid psychiatric disorder (as determined by investigators - e.g., schizophrenia or bipolar disorder) and/or psychosis at the time of study enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rivermead Post-Concussion Symptoms Questionnaire | Baseline, immediately before the first iTBS treatment
  A validated measure of subjective global PCS symptoms
Rivermead Post-Concussion Symptoms Questionnaire | 5 days
  A validated measure of subjective global PCS symptoms
Rivermead Post-Concussion Symptoms Questionnaire | 1 month post-treatment
  A validated measure of subjective global PCS symptoms

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | Baseline, post treatment day 5, and Study endpoint
  Montgomery-Åsberg Depression Rating Scale is a widely used clinician-rated measure of depressive severity
Repeatable Battery for the Assessment of Neuropsychological Status | Baseline and post treatment 1 month
  Repeatable Battery for the Assessment of Neuropsychological Status is a brief, individually administered battery to measure cognitive decline or improvement
The Behavior Rating Inventory of Executive Function | Baseline, post treatment day 5, and post treatment 1 month
  The Behavior Rating Inventory of Executive Function-A is a standardized measure that captures views of an adult's executive functions or self-regulation in his or her everyday environment.
Headache Impact Test | Baseline and post treatment 1 month
  Headache Impact Test is a tool used to measure the impact headaches have on one's ability to function on the job, at school, at home and in social situations.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided